CLINICAL TRIAL: NCT00754390
Title: Effects of Calcium and Phytate on Zinc Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: GFHNRC042
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2009-06-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Dietary Zinc Absorption
Keywords: dietary zinc absorption; dietary phytic acid; dietary calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Study (Experimental): Participants consumed 4 experimental diets for 4 weeks each in randomized order
  Interventions: Dietary Supplement: Moderate Calcium, Low phytate Diet; Dietary Supplement: Moderate Calcium, High Phytate Diet; Dietary Supplement: High Calcium, Low Phytate Diet; Dietary Supplement: High Calcium, High Phytate Diet

INTERVENTIONS:
Dietary Supplement: Moderate Calcium, Low phytate Diet — Participants consumed diet containing 700 milligrams calcium and 440 milligrams of phytate for 4 weeks
Dietary Supplement: Moderate Calcium, High Phytate Diet — Participants consumed diet containing 700 milligrams calcium and 1800 milligrams of phytate for 4 weeks
Dietary Supplement: High Calcium, Low Phytate Diet — Participants consumed diet containing 1900 milligrams calcium and 440 milligrams of phytate for 4 weeks
Dietary Supplement: High Calcium, High Phytate Diet — Participants consumed diet containing 1900 milligrams calcium and 1800 milligrams of phytate for 4 weeks

SUMMARY:
This study is determine the effects of dietary calcium and phytate on zinc absorption.

DETAILED DESCRIPTION:
Zinc absorption is tested from 2 days of consuming each of four diets with zinc-65 isotope, followed by retention monitoring in a whole body scintillation counter for 4 weeks. All four 4 experimental diets are tested with each subject, in randomized order, for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Average weight for height

Exclusion Criteria:

* Medications other than birth control pills or hormone replacement therapy,
* Pregnancy within last 6 months

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet R Hunt, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- United States Department of Agriculture Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited by the United States Department of Agriculture (USDA) Grand Forks Human Nutrition Research Center to participate in an out-patient feeding study in Grand Forks, North Dakota
Pre-assignment Details: 205 participants applied, 157 were eligible, 27 accepted invitation to attend an information meeting, 10 started study, 7 of the alternates joined study as original participants withdrew or were discharged.
Groups:
- Calcium and Phytate Interactions: Subjects consumed 4 test meals (Moderate Calcium (Ca),Low Phytate; Moderate Ca,High Phytate; High Ca,Low Phytate; High Ca,High Phytate) in random order
Period: Ca/Phytate Test Meal 1 (Randomized)
Arm/Group | Calcium and Phytate Interactions
Started | 17
Completed | 12
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 2
Period: Ca/Phytate Test Meal 2 (Randomized)
Arm/Group | Calcium and Phytate Interactions
Started | 12
Completed | 12
Not Completed | 0
Period: Ca/Phytate Test Meal 3 (Randomized)
Arm/Group | Calcium and Phytate Interactions
Started | 12
Completed | 11
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Ca/Phytate Test Meal 4 (Randomized)
Arm/Group | Calcium and Phytate Interactions
Started | 11
Completed | 10
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all subjects randomized to the 4 treatments. Treatments were assigned in randomized order so the number of subjects starting the study does not equal the starting number for a given treatment
Arm/Group | Entire Study Population
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Zinc Absorption
Description: Retention of Zinc-65 was monitored for 28 days by whole body scintillation counting. The percentage of Zinc-65 absorbed was estimated from the y-intercept of the linear portion of a semilogarithmic retention plot of percent Zinc-65 retained versus time
Time Frame: 16 weeks
Population: Analysis restricted to women who completed all 4 treatment periods
Measure: Mean (Standard Error); unit: Percentage of Zinc-65 absorbed
Groups:
- Moderate Calcium, Low Phytate Diet: Two days of radiolabelled diet containing 700 milligrams of Calcium per day and 440 milligrams of phytate per day
- Moderate Calcium, High Phytate Diet: Two days of radiolabelled diet containing 700 milligrams of Calcium per day and 1800 milligrams of phytate per day
- High Calcium, Low Phytate Diet: Two days of radiolabelled diet containing 1900 milligrams of Calcium per day and 440 milligrams of phytate per day
- High Calcium, High Phytate Diet: Two days of radiolabelled diet containing 1900 milligrams of Calcium per day and 1800 milligrams of phytate per day
Arm/Group | Moderate Calcium, Low Phytate Diet | Moderate Calcium, High Phytate Diet | High Calcium, Low Phytate Diet | High Calcium, High Phytate Diet
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage of Zinc-65 absorbed | 32.8 (2.3) | 26.9 (2.4) | 39.4 (2.4) | 26.2 (2.3)
Statistical Analysis 1: Comparison: Moderate Calcium, Low Phytate Diet vs Moderate Calcium, High Phytate Diet vs High Calcium, Low Phytate Diet vs High Calcium, High Phytate Diet; Two-way mixed model analysis of variance was used to test for main effect of dietary calcium and phytate and their interaction. Null Hypothesis: Dietary calcium does not affect zinc absorption; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis
Statistical Analysis 2: Comparison: Moderate Calcium, Low Phytate Diet vs Moderate Calcium, High Phytate Diet vs High Calcium, Low Phytate Diet vs High Calcium, High Phytate Diet; Two-way mixed model analysis of variance was used to test for main effect of dietary calcium and phytate and their interaction. Null Hypothesis: Dietary Phytate does not affect zinc absorption; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis
Statistical Analysis 3: Comparison: Moderate Calcium, Low Phytate Diet vs Moderate Calcium, High Phytate Diet vs High Calcium, Low Phytate Diet vs High Calcium, High Phytate Diet; Two-way mixed model analysis of variance was used to test for main effect of dietary calcium and phytate and their interaction. Null Hypothesis: Dietary calcium and dietary phytate do not affect zinc absorption. Eight women were required to detect a difference in zinc absorption of 7 percentage points with a power of 90%, alpha level of 0.05; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Overall Study: Participants consumed 4 dietary treatments in randomized order
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes